CLINICAL TRIAL: NCT04772430
Title: Zonguldak Bulent Ecevit University
Brief Title: "The Effect of Snow Globe Used in Infancy Vaccination Applications on Pain Level."
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zonguldak Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, Betul Akkoc, Zonguldak Bulent Ecevit University, Zonguldak Bulent Ecevit University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 12102020100140
Record Dates: First submitted 2021-02-22; First posted 2021-02-26 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Pain
Keywords: pain; immunization; diverting attention; infancy
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): The baby whose height and weight measurements will be taken will be taken to the stretcher, and the vaccine will be administered after the pain score is measured before the procedure. Pain scores will be recorded during and after the procedure
- Experimental group (Experimental): The baby whose height and weight measurements will be taken will be taken to the stretcher, after the pain score is measured before the procedure, the snow globe will be operated and the vaccine will be applied. The snow globe will continue to work until the application is completed. Pain scores will be recorded during and after the procedure.
  Interventions: Radiation: snow globe

INTERVENTIONS:
Radiation: snow globe — Control group; The baby whose height and weight measurements will be taken will be taken to the stretcher, and the vaccine will be administered after the pain score is measured before the procedure. Pain scores will be recorded during and after the procedure.
  Experimental group; The baby whose height and weight measurements will be taken will be taken to the stretcher, after the pain score is measured before the procedure, the snow globe will be operated and the vaccine will be applied. The snow globe will continue to work until the application is completed. Pain scores will be recorded during and after the procedure.
  Arms: Experimental group

SUMMARY:
The aim of this research is to determine the effect of the snow globe, which is used as a method of diverting attention, to the perception of pain that develops during the application of vaccines in infants between 2-6 months of age.

DETAILED DESCRIPTION:
Atraumatic care philosophy developed by Donna Wong; it is a principle of therapeutic care aimed at minimizing or eliminating the physical and psychological problems experienced by the child and his/her family. Pediatric nurse; it is obliged to offer atraumatic care by ensuring the cooperation of the child and his/her family, reducing pain and controlling stressors.

In accordance with the principles of atraumatic care; limitation of painful initiatives to prevent or reduce physical stress sources, regulation of environmental conditions, use of pharmacological and nonpharmamological pain removal methods in the presence of pain; promoting family-centered care in order to ensure the unity of children and family members; informing the child and his family about care to ensure the development of a sense of control, resting recommendations on care, establishing a daily care program.

The American Pain Association considers pain the fifth life finding. Studies show that all babies, including preterm babies, suffer pain and can distinguish pain from other sensory experiences. Controlling pain in children is multidisciplinary team work. It makes the nurse different from other team members in the control of pain and ensures that she is in an indispensable position; the nurse spends a long time with children, learns about the child's previous pain experiences and methods of coping with pain and benefits from coping methods when necessary, teaching the child and his family strategies to cope with pain, guiding them, applying planned treatment, monitoring their effects, results and empathizing, in short, being able to practice the nursing process.

Children who are often subjected to painful invasive interventions from the newborn period; however, they have a structure that requires the consideration of their level of development, cognitive and communicative skills, previous experiences of pain. According to the American Academy of Pediatrics , newborns and children are exposed to a total of 24 injections due to vaccination in the first 2 years of their life. In Turkey, the total number of injections for routine vaccination of children up to 2 years of age is 18. The negative effects of pain, which cannot be managed effectively, in physiological and psychological dimensions can occur even years later. The pain and stress experienced with deterioration in the clinical condition of newborns brings many complications.

Pain in children is more difficult to assess than in adults. The perception of pain in children, age, gender, family reactions to pain, previous experiences, insomnia, fatigue, fear, sadness, anger, being in an unpleasant environment can affect.

Conditions caused by pain include short-term changes such as respiratory irregularity, hypoxemia, fading or redness, blood pressure changes, increased heart rate and oxygen consumption, enlargement of pupils, as well as permanent, structural and functional (endocrine, behavior and immune system) changes. It negatively affects the behavior, family infant interaction, diet and clinical course of babies who warn of long-term and frequent pain, as well as prevents the baby's adaptation to the outside world. Repeated painful interventions can lead to neurotoxia and lead to deterioration in social cohesion, anxiety, change in pain sensitivity, stress disorders, hyperactivity/attention deprivation in the future. That's why the American Pain Society (APS) and the American Academy Of Pediatrics (AAP) recommend minimizing pain and anxiety due to procedures. The high number of vaccines for children and infants and the psychological traumas caused by the pain caused by the vaccines make it mandatory to intervene in the pain that occurs during vaccination and are one of the ethical issues

Research shows that nurses do not make adequate pain assessments and do not use nonpharmamological methods effectively. Nonpharmaciological pain methods, which are effective in consequential or alone, can also be used in the elimination of pain, among the non-pharmacological methods such as hot cold application, diverting attention, listening to music, balloon blowing, reading books, watching movies, vibration, transcutaneous electrical nerve stimulation (transcutaneous electrical nerve stimulation) application.

Divert attention; it is a non-drug method that is often used in the management of pain in children. It removes the perception of pain by focusing the individual's attention away from pain and in another focus. More work is needed to improve pain management in children and illuminate optimal pain management and strategies that take into account children-specific needs

ELIGIBILITY:
Inclusion Criteria:

* Being registered at Bartın Family Health Center
* Being in the age range of 2-6 months
* Having parental consent
* Does not have a congenital or chronic health problem,
* Not taking an analgesic drug in the last 4 hours,
* Infants of families who have accepted to participate in the study and signed the informed consent form will be included in the study

Exclusion Criteria:

* Being aged between 0-1 months and over 6 months,
* No parental consent,
* Using analgesics in the last 4 hours,
* The child has a congenital or chronic health problem

Ages: 2 Months to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2021-04-01 (Estimated)

PRIMARY OUTCOMES:
Face, Legs, Activity, Cry, Consolability (FLACC) Behavioral Pain Scale | 2-6 months
  Flacc pain scale score is obtained by evaluating in five categories as facial expression, leg movements, activity, crying and consolingness. By giving 0, 1, or 2 points for each category, the total score between 0 and 10 is reached. As the pain intensity increases, the total score increases, as the pain intensity decreases, the total score decreases

SECONDARY OUTCOMES:
Heart rate | 2-6 months
  heart rate of the babies were recorded using a pulse oximeter placed on the right or left foot or hand of each baby before the invention. heart rate levels were recorded during and after vaccination .
oxygen saturation | 2-6 months
  oxygen saturation of the babies were recorded using a pulse oximeter placed on the right or left foot or hand of each baby before the intervention. oxygen saturation levels were recirded during anda after vaccination
crying duration of babies | 2-6 months
  the crying time was expressed in seconds. The crying time is measured and recorded with the stopwatch before and after the procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- Betül Akkoç, Merkez, Bartın, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No